CLINICAL TRIAL: NCT04539990
Title: A Behavioral Intervention for Ameliorating Sleep Problems in Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sor 0266-20 ctil
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Autism; Autism Spectrum Disorder; Sleep
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Sleep Treatment (Experimental): Parents of children with autism will come to two group meetings (up to 5 families in each group) where they will be receive information regarding sleep hygiene and behavioral techniques for reducing sleep onset delays and night awakenings. The program will last 8 weeks. Meetings will be held on week 1 and week 3. In addition parents will receive a weekly phone call where they will be asked about their ability to implement the behavioral techniques.
  Sleep of the children will be measured using questionnaires, sleep diaries and with a Fitbit sensor before and after the program.
  Interventions: Behavioral: Behavioral treatment for sleep difficulties

INTERVENTIONS:
Behavioral: Behavioral treatment for sleep difficulties — This intervention is mediated by the parents. Parents are educated regarding sleep hygiene and instructed to follow simple rules which create a reliable evening routine and reduce exposure to stimulating factors that delay sleep onset (e.g., caffeine or exercise). In addition, parents are asked to initiate a "fading" behavioral protocol whereby they teach their child to fall asleep independently, with less parental attention. This requires parents to limit their interaction with their child after the children are put to bed so as not to interfere with sleep onset. This includes limiting conversations and lying in bed with the child. This behavioral approach is applied gradually and is expected to reduce the time it takes children to fall asleep.

SUMMARY:
The present study will test the effectiveness of a behavioral intervention program that targets sleep problems in 1.5-5-year-old children with ASD. Sleep patterns will be measured using questionnaires and sleep diaries that will be completed by the parents as well as by Fitbit sensors that will be placed on the child's wrist or back of the arm. The study will also explore whether specific child (e.g., severity of cognitive abilities) or parent characteristics (e.g., parent stress levels) impact the effectiveness of the intervention. In addition, we will examine whether changes in sleep disturbances are associated with changes in the family's quality of life.

ELIGIBILITY:
Inclusion Criteria:

Parents of 1.5-5-year-old children with autism will be asked to fill the Child Sleep Habits Questionnaire (CSHQ). Those who report high scores on the following 3 CSHQ subscales will be invited to participate: bedtime resistance, sleep onset delay, and night-wakings.

Exclusion Criteria:

None

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Child Sleep Habits Questionnaire | 8 weeks after program begins
  Parent questionnaire regarding sleep habits of their child
Night time sleep as measured by Fitbit sensor | 8 weeks after program begins
  Sensor is placed on the arm of the child for 5 days and measures sleep